CLINICAL TRIAL: NCT01336426
Title: Clinical Trial for Evaluation of Vermillion's Blood Test to Predict the Probability of Peripheral Artery Disease
Acronym: PAD-001
Status: Completed | Type: Observational
Sponsor: Vermillion, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: PAD-001
Record Dates: First submitted 2011-04-06; First posted 2011-04-15 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma and Frozen Red Blood Cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose

This study is to verify and validate PAD1 as a qualitative serum test which will combine the results of multiple assays into a single numeric result, to be determined by evaluation of the study data.

PAD1 is an automated software device (PADCalc) that incorporates specific and multiple biomarker values found in human blood, and generates a score (PAD1 score) using a fixed formula implemented within the PADCalc software. The PAD1 score is a result with a high or low probability of PAD.

PAD1 will be submitted to FDA as a 510(k) for in vitro diagnostic use in conjunction with clinical assessment, based on factors such as age, diabetes, smoking, and vascular laboratory tests (including the ABI), as an aid towards further evaluation of patients who meet the enrollment eligilbility criteria.

Eligibility It is indicated for women and men considered at risk for PAD who meet the following criteria: a history of smoking and/or diabetes and are age 50 years or older, or 70 years of age or older. PAD1 is an aid to further assess the likelihood of the presence of PAD when used in conjunction with clinical assessment and vascular laboratory tests.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) affects 8 to 12 million individuals in the United States and is also prevalent in Europe and Asia. A regional pilot study of community screening for PAD demonstrated that patient awareness of a PAD diagnosis was low, and was associated with atherosclerosis risk factors, antiplatelet therapy, and claudication treatment intensity. PAD has not emerged as a focus of public health efforts to improve quality of life, nor to decrease the associated cardiovascular ischemic risk. Smoking, diabetes, and age are the strongest risk factors for PAD. Smokers have a 2 to 6-fold increased likelihood of having PAD, and the risk of PAD increases in a dose-dependent manner with the duration and amount of smoking. Diabetes confers a 2 to 4-fold increased risk of having PAD. The prevalence of PAD increases as a function of age. Criqui et al showed that the prevalence of PAD in individuals under 60 years of age was about 2.5%, whereas the prevalence increased to over 20% in individuals over 75 years of age.

A study in smokers and diabetics 50 years of age or older, and in all those 70 years of age or older, identified in an outpatient, primary care clinic setting has shown that the prevalence is 29%. About half of the cases found were newly-identified PAD patients. Further, while 83% of those with a prior diagnosis of PAD were aware of their condition, only 49% of the primary-care physicians were aware that their patients had a diagnosis of PAD. Another study examined internal medicine physicians' approaches to PAD and found that only 37% reported taking histories for claudication, and only 26% evaluated the foot for ulcers.

PAD is as prevalent in women as in men. When symptomatic, PAD causes limb discomfort, tiredness, heaviness, cramping, or pain brought on by exertion and relieved by rest (i.e., intermittent claudication) and reduces functional capacity and quality of life. Classic claudication is only noted by 10-30% of patients and atypical leg discomfort occurs in 20-40%. Up to 50% of patients are asymptomatic. PAD1 is an in vitro diagnostic that provides a PAD1 score derived from multiple biomarkers in human plasma, serum, or whole blood, which predicts a low or high probability of the presence of PAD in patients at risk for PAD. A positive PAD1 score(above the cutoff), indicating a higher risk for PAD than expected in the general population, would then guide the physician to more aggressively determine the presence of PAD.

The preliminary studies have shown an association of four proposed biomarkers with ABI, and have demonstrated the construction of a PAD risk algorithm. This study is powered to test each of the four biomarkers and their interactions and develop the PAD1 risk score in the intended use population.

ELIGIBILITY:
Inclusion Criteria:

Subject is one or more of the following:

* ≥50 years old and subject-reported current or former history (<10 years) of smoking for a minimum of 10 pack years.
* ≥50 years old and history of type 2 diabetes (meeting American Diabetes Association criteria) as documented in the medical record, or use of diabetes medications or diabetes-specific diet.
* ≥70 years old. 2. Subject provides written informed consent to participate in this study. 3. Subject agrees to de-identified biorepository storage of own processed blood sample for future testing.

Exclusion Criteria:

1. Significant hepatic or renal insufficiency, including either of the following:

   * Renal insufficiency or renal failure within the past 6 months, or creatinine >2.5 mg/dL within the past 6 months (if results available), or currently on dialysis.
   * Severe liver disease or any chronic hepatitis within the past 6 months, or AST and ALT >3xULN (upper limit of normal), or bilirubin >2xULN within the past 6 months (if results available).
2. Active viral or bacterial infection or subject is currently taking an antibiotic or antiviral agent.
3. Active inflammatory condition requiring treatment with systemic steroids or immune modulating therapy within the past 6 months.
4. Active malignancy that requires active anti-neoplastic therapy (stable basal cell skin cancer is allowed; cancer being treated solely with hormonal therapy is allowed).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that meet the inclusion/exclusion criteria from 10 primary care sites.
Sampling Method: Probability Sample
Enrollment: 1033 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
PAD1 will identify individuals with a higher risk of PAD. | 1 month
  PAD1 will identify individuals with a higher risk of PAD in an at-risk population of individuals 70 years of age or older, or smokers and/or diabetics 50 years of age or older.

SECONDARY OUTCOMES:
To demonstrate that PAD1 has predictive value for PAD when used as a combination result. | 1 month
  To demonstrate that PAD1 has predictive value for PAD in combination with:
  * The Framingham Risk Score
  * The 5-Symptom Questionnaire for prediction of PAD (5-Q Sx)

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Fung, MD. PhD., Study Director — Vermillion, Inc.
Locations (10):
- United States (10):
  - Coastal Clinical Research, Mobile, Alabama
  - Apex Research Institute, Santa Ana, California
  - Radiant Research, Santa Rosa, California
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Lovelace Scientific Research, Albuquerque, New Mexico
  - Radiant Research, Columbus, Ohio
  - Omega Clinical Research, Warwick, Rhode Island
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - National Clinical Research, Inc., Richmond, Virginia